CLINICAL TRIAL: NCT02679391
Title: The Outcome of Abdominoplasty After Massive Weight Loss; Comparison of Results From Plastic and General Surgical Units - a Retrospective Cohort Study
Brief Title: The Outcome of Abdominoplasty After Massive Weight Loss
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, prof. Ulf Gunnarsson, Professor, Karolinska Institutet
Other Study IDs: ES2012/1997-31/4
Record Dates: First submitted 2016-01-27; First posted 2016-02-10 (Estimated); Last update posted 2016-02-10 (Estimated); Status verified 2016-02

CONDITIONS: Weight Loss
Keywords: Abdominoplasty; Early complications; Guidelines; Sequelae; bariatric patients
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- A: 69 consecutive operated patients by general surgeons at Capio S:t Görans Hospital 2011. All post weight loss. , 96% female, BMI by the time of operation 26, mean age 41 (SD 9.5). Their mean weight loss in BMI units: 17.8 (SD 5.12).
- B: 70 consecutive operated patients by plastic surgeons at Karolinska University Hospital 2010-2012. All post weight loss. 86% female, BMI by the time of oepration 26, mean age 38.6 (SD 11.4). Their mean weight loss in BMI units: 17.4 (SD 4.8).
- C: 70 consecutive operated patients by general surgeons at Capio S:t Görans Hospital 2013-2014. All post weight loss. 90% female, BMI by the time of operation 26, mean age 46.8 (SD 10.1). Their mean weight loss in BMI units: 16.3 (SD 5.11)

SUMMARY:
The primary aim of this study is to compare early surgical complications after abdominoplasty performed by plastic and general surgeons. Secondary aims were to assess whether specific guidelines might have impact on the rate of complications. The hypothesis is that general surgeons have more complications.

DETAILED DESCRIPTION:
Bariatric surgery has gained widespread acceptance and 6,800 patients are yearly operated in Sweden. Approximately 30 % of these patients require abdominoplasties for functional disabilities being a total of 2,300 patients. Today the plastic surgeons of the departments of Plastic and Reconstructive Surgery do not have the capacity to accommodate this demand. A Department of General Surgery started to perform abdominoplasties.

This is a retrospective cohort study. Charts were retrieved from 69 consecutive patients operated by general surgeons at Capio S:t Görans Hospital, Stockholm, Sweden (group A) from 13th of May to 19th of December 2011. Charts from 70 consecutive patients operated by plastic surgeons at the Department of Plastic and Reconstructive Surgery, Karolinska University Hospital, Stockholm, Sweden (group B) were studied from 14th of January 2010 to 7th of December 2012. Collected data consist of patient demographics, operation methods, and complications observed at 30 days' follow-up. The outcome of a third group of about 70 patients operated between 22th of January 2013 to 3th of June 2014 at S:t Görans Hospital (group C) are compared to the outcome of groups B and A. Guidelines for the surgical technique as well as pre-and postoperative care were refined between the operations of group A and C.

Statistics Anova and regression analysis will be applied. And for dichotomous data Chi-Square test and Fischers exact test will be calculated. Power was calculated with the test of proportion for two independent groups and 5 per cent significance.

ELIGIBILITY:
Inclusion Criteria:

* Abdominal skin ptosis > 3 cm
* Weight stability > 6 months
* Smoke free > 6 weeks prior to surgery
* BMI ≤28 or a significant weight reduction equivalent to 80 per cent of excess weight

Exclusion Criteria:

* Weight instability
* Smoking
* BMI >35
* Psychological imbalance or psychiatric non-treated diseases
* Advanced cardio-vascular diseases

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients that were accepted for abdominoplasties after massive weight loss in accordance with the inclusion and exclusion criterias. Consecutively operated.
Sampling Method: Probability Sample
Enrollment: 209 (Actual)
Dates: Start 2010-01; Primary Completion 2014-06 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Comparing postoperative complications after abdominoplasty performed by plastic and general surgeons, where the dichotomous variables are evaluated. | 1 month follow up
  Dichotomous data yes/no collected in Excel from the charts. The complications are: wound infection, wound dehiscence, seromas, bleeding, transfusions, tissue necrosis, systemic disorder, lung embolism, Deep venous thrombolism, reoperation, hospital stay over 2 Days and Patients with no adverse effect.

SECONDARY OUTCOMES:
Secondary aims were to assess whether specific guidelines might have impact on the rate of complications, concerning the same complications as mentioned in the primary outcome. | 4 years
  Between two of the cohorts new guidelines was introduced, and the same dichotomous data (yes/no) was collected and with logistic regression analyzed to assess if the applied guidelines made any effect on the complications. The guidelines, if followed, was yes/no.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Brännström, MD. PhD, Study Director — Karolinska Institutet

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Swedenhammar E, Stark B, Hallstrand AH, Ehrstrom M, Gahm J. Surgical Training and Standardised Management Guidelines Improved the 30-Day Complication Rate After Abdominoplasty for Massive Weight Loss. World J Surg. 2018 Jun;42(6):1647-1654. doi: 10.1007/s00268-017-4341-8. PMID 29185021